CLINICAL TRIAL: NCT03659721
Title: The Effects of Family Clinic and Municipality (FACAM)
Brief Title: The Effects of Family Clinic and Municipality
Acronym: FACAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: Odense University Hospital (Other); Syddansk Universitet (Unknown); Odense Patient Data Explorative Network (Other); Odense Kommune (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VIVE 100750-751
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: At-risk Pregnant Women
Keywords: Pregnant; Infant; Parent; Family; Mother; Support

STUDY DESIGN:
Intervention Model Description: The study is a prospective randomized controlled trial with two study arms: intervention (FACAM) and care as usual (CAU). Pregnant women are randomized to receive either FACAM or CAU.
Who Masked: Investigator, Outcomes Assessor
Masking Description: As the participants are offered extra support as the intervention neither participants nor care providers can be blinded. Outcome assessor and data analyst will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACAM (Experimental): Intervention participants are assigned a support person (health nurse or a family therapist) who will offer support to the family until the child starts school at age 6. Intensity is up to 37 hours the first year followed by up to 10 hours of support each of the following years. The support person will offer individualized support to the family depending on the needs of the family. The support person will attend midwife consultations and help the pregnant woman to attend consultations with e.g. GP, midwife, or social worker. All intervention participants will also receive either an individual or group-based (COS-P)attachment based intervention during pregnancy and the first months of the child's life.
  Interventions: Behavioral: FACAM; Behavioral: COS-P
- Care as Usual (Active Comparator): Families in the control group receive the usual care that is offered to families in the target group. This includes consultations with e.g. a midwife, social worker, medical doctor, and health visitor. If needed, CAU families can receive e.g. extra home visits or family therapy.
  Interventions: Behavioral: Care as Usual

INTERVENTIONS:
Behavioral: FACAM — Support person
  Arms: FACAM
Behavioral: Care as Usual — Usual care
  Arms: Care as Usual
Behavioral: COS-P — Attachment based therapy
  Arms: FACAM

SUMMARY:
This trial is a randomized controlled trial with the aim is to assess the effectiveness of Family Clinic and Municipality (FACAM) to improve mother-child relationship, maternal health, maternal mental health, and the development and well-being of the child.

DETAILED DESCRIPTION:
Pregnant women who struggle with psychosocial challenges during pregnancy have a higher risk of preterm birth, giving birth to a child with low birth weight and a higher risk of complications during pregnancy both for mother and child. An early and coordinated intervention to reduce inequality in health may be important for this group of vulnerable women.

The FACAM intervention is developed in Odense with the aim of reducing inequality in health by giving vulnerable pregnant women and their children the best possible start in life by offering an interdisciplinary coordinated support. The support will be offered by Odense municipality, the family clinic (Familieambulatoriet), and local voluntary organizations.

The aim of the trial is to assess the effectiveness of FACAM to improve mother-child relationship, maternal health, maternal mental health, and the development and well-being of the child.

The study is a Randomized Controlled Trial (RCT). A total of 320 pregnant women will be randomized to FACAM or Care as Usual.

Participants are pregnant women categorized as antenatal care group 3 or 4, living in Odense and with a referral to Familieambulatoriet, OUH. Participants must be able to fill out questionnaires in Danish or English.

Data will be collected at baseline (pregnancy), and when the child is 3 and 12 months old.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women admitted to the Familieambulatorium, and living in Odense municipality
* Antenatal care group 3 or 4 according to the Danish health authorities' recommendations

Exclusion Criteria:

* Life-threatening illness in parent or child
* Not able to fill out questionnaires in Danish or English
* Child in out of home care after birth
* Pregnancy with twins
* Previous participation in the FACAM project

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants must be pregnant women
Enrollment: 332 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Maternal sensitivity | at child age 12 months
  Maternal sensitivity measured by the CIB (Coding Interactive Behavior)

SECONDARY OUTCOMES:
Maternal Sensitivity | at child age 3 months
  Maternal sensitivity measured by the CIB (Coding Interactive Behavior)
Coding interactive bahavior (CIB) | child age 3 and 12 months
  Parent child relationship Subscales: Intrusiveness, Limit setting, Involvement, Withdrawal, Reciprocity, Negative states
Ages and Stages Questionnaire-Social Emotional 2 (ASQ:SE-2) | child age 3 and 12 months
  Child social-emotional Development Total score range 0-150 ( 3 months 15 items), 0-260 (12 months 26 items). Low score is better.
Edinburgh Postnatal depression Scale (EPDS) | child age 3 and 12 months
  Depression Total score range 0-30. Low score is better
Warwick-Edinburgh Mental Well-being Scale | child age 3 and 12 months
  Maternal mental Health 7 items. A total score i calculated by summing the 7 items and converting the raw score according to a published conversion table. Raw score range 7- 35. Converted score range 7-35. High is better outcome.
Prenatal Parental reflective functioning questionnaire (P-PRFQ) | Baseline
  Parental reflective functioning for pregnant women. Total score range 14-98. Higher score is better. Three subscales:
  Opacity of mental states (4 items), reflecting on the fetus-baby (3 items) and Dynamic of mental states (5 items)
Parental reflective functioning questionnaire (PRFQ-1) | child age 12 months
  Parental reflective functioning Three subscales score range 6-42: Pre-Mentalizing Modes (PRFQ-PM) 6 items. low score is better. Certainty about Mental States (PRFQ-CMS) 6 items high score is better. Interest and curiosity in mental states PRFQ-IC 6 items high score is better.
Parental Stress Scale (PSS) | Cild age 3 and 12 months
  Parental stress Total score range 18-90 low score is better
Ages and Stages Questionnaire 3 (ASQ:3) | child age 3 months
  Child development
Activities with child | child age 12 months
  Singing and reading Total score range 0-70. High score is better.
Being a Mother (BAM-13) | child age 3 and 12 months
  Maternal confidence. Total score range 0-39. Low score is better
Hospital Anxiety and Depression Scale (HADS) | Baseline, 3 and 12 months
  Two subscales Anxiety (range 0-21 low score is better) and depression (range 0-21 low score is better)
Experiences in Close Relationship Scale-Short Form (ECR-S) | Baseline
  Two subscales Anxiety (range 1-42 low score is better) and Avoidance (range 1-42 low score is better)

CONTACTS AND LOCATIONS:
Overall Officials: Maiken Pontoppidan, PhD, Principal Investigator — VIVE
Locations (2):
- Denmark (2):
  - VIVE - The Danish Centre of Social Science Research, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol and analysis plan will be available

REFERENCES:
- [Derived] Pontoppidan M, Nygaard L, Thorsager M, Friis-Hansen M, Davis D, Nohr EA. The FACAM study: protocol for a randomized controlled study of an early interdisciplinary intervention to support women in vulnerable positions through pregnancy and the first 5 years of motherhood. Trials. 2022 Jan 24;23(1):73. doi: 10.1186/s13063-022-06022-4. PMID 35073975